CLINICAL TRIAL: NCT02120131
Title: Trapezoidal Flap Versus Envelope Flap in Impacted Mandibular Third Molar Extraction
Brief Title: Trapezoidal Flap vs. Envelope Flap in Mandibular Third Molar Extraction.
Status: Completed | Type: Observational
Sponsor: University of Firenze and Siena, Napoli, Italy (Other)
Responsible Party: Principal Investigator, nicola baldini, oral surgeon, University of Firenze and Siena, Napoli, Italy
Other Study IDs: pcttm
Record Dates: First submitted 2014-04-15; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Impacted Third Molar Tooth
Keywords: third molar surgery, periodontal probing depth , flap design

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- test envelope: envelope flap
- control, trapezodal: standard incision

SUMMARY:
the purpose of this study was to test the effectiveness of the envelope flap compared to trapezoidal flap in impacted mandibular third molar extractions.

DETAILED DESCRIPTION:
a sample of 50 patients requiring mandibular third molar extraction was selected for the study. Healthy patients with mild symptoms of pericoronitis affecting at least 1 mandibular third molar were included in the study. A total number of 52 consecutive cases of mandibular third molar surgical extractions were performed using either a trapezoidal flap or an envelope flap. The choice of the flap was randomized. The following parameters were recorded: Probing Pocket Depth, Clinical Attachment Level, Bleeding on Probing, Full Mouth Plaque Score, Full Mouth Bleeding Score, total time for the surgical intervention, age of the patient, type of inclusion, ostectomy. All the patients received a questionnaire to evaluate the post-intervention discomfort (swelling, pain, number of pain-killers, bleeding). Periodontal parameters were checked at 6-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* third molar impaction
* mild symptoms of pericoronitis

Exclusion Criteria:

* systemic diseases
* cigarettes smoking
* history of irradiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: a sample of 50 patients requiring mandibular third molar extracion was selected for the study. Healthy patients with mild symptoms of pericoronitis affecting at least 1 mandibular third molar were included in the study
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
change from baseline on the periodontal status of adjacent second molar | 6 months

SECONDARY OUTCOMES:
post surgical complication | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: nicola nb baldini, oral surgeon, Principal Investigator — tuscan scool of dental medicine of florence and siena
Locations (1):
- Tuscan School of Dentistry, Siena, Siena, Italy